CLINICAL TRIAL: NCT02949258
Title: A Phase II Study of Neoadjuvant Chemotherapy With SEEOX Regimen Via Intra-arterial and Intravenous Administration Followed by Surgery for Borrmann Type 4 Gastric Cancer
Brief Title: Neoadjuvant Chemotherapy With SEEOX Regimen for Borrmann Type 4 Gastric Cancer
Acronym: NCT-B4
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Li Guoli, Professor, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4-2016-LGL
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Stomach Neoplasms; Gastric Cancer
Keywords: gastric cancer; Borrmann type 4; Neoadjuvant chemotherapy; Intra-arterial administration
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Etoposide; Epirubicin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SEEOX group (Experimental): A three-cycle neoadjuvant chemotherapy will be performed in all cases. In every cycle, oxaliplatin 150 mg, etoposide 100 mg and epirubicin 50 mg will be administered from the celiac artery on day 1. Oral S-1 120 mg per day will be given for days 1-14. The second cycle will be scheduled following a 1-week rest after the first cycle.After two courses of neoadjuvant chemotherapy, patients will be reevaluated and receive curative or palliative resection or exploratory laparotomy within 14 days after completing the second course of chemotherapy.
  Interventions: Drug: oxaliplatin; Drug: etoposide; Drug: epirubicin; Drug: S1

INTERVENTIONS:
Drug: oxaliplatin — oxaliplatin 150 mg will be administered from the celiac artery on day 1 of every cycle in all cases
Drug: etoposide — etoposide 100 mg will be administered from the celiac artery on day 1 of every cycle in all cases
Drug: epirubicin — epirubicin 30 mg will be administered from the celiac artery on day 1 of every cycle in all cases
Drug: S1 — Oral S-1 120 mg per day will be administered on days 1-14 of every cycle in all cases

SUMMARY:
Scirrhous gastric cancer, also known as linitis plastic or Borrmann type 4, is an aggressive tumor with an extremely poor prognosis. Aggressive surgical procedures and adjuvant chemotherapies have not improved the survival rate. The purpose of this study is to determine whether neoadjuvant Chemotherapy with SEEOX regimen via intra-arterial and intravenous administration are effective in the treatment of Borrmann type 4 gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer patients who diagnosed as Borrmann type 4 would be included in this study.They would receive 3 cycles of neoadjuvant chemotherapy with SEEOX regimen via combined intra-arterial and intravenous administration. The treatment schedule consisted of 3 courses (each, 2-week administration and 1-week withdrawal) of intra-arterial administration of oxaliplatin (150mg), etoposide (100mg) and epirubicin(30mg) by Seldinger method on day 1 and oral S-1(120mg) on days 1-14, followed by radical surgery.The efficacy and toxicity of SEEOX regimen would be examined.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed gastric adenocarcinoma;
* males or females, aged 30-70 years;
* gastroscopy and abdominal computed tomography (CT) scan-confirmed typical scirrhous gastric cancer (without definitive ulceration) that invaded more than half of the stomach;
* no peritoneal metastasis confirmed by laparoscopic exploration and with cytological examination of peritoneal washing of the Douglas pouch;
* eastern Cooperative Oncology Group performance status of 0 or 1;
* no serious concomitant diseases that make survival period < 3 years;
* no prior anti-tumor therapy;
* have signed informed consent before the beginning of treatment.

Exclusion Criteria:

* patients can not bear surgical procedure;
* pregnant or lactating women;
* previous cytotoxic chemotherapy, radiotherapy or immunotherapy;
* with peritoneal metastasis or distant metastasis;
* history of another malignancy within the last five years;
* history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the Investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake;
* clinically significant (i.e. active) cardiac disease e.g. symptomatic coronary artery disease, New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication or myocardial infarction within the last 12 months;
* organ allografts requiring immunosuppressive therapy;
* serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease;
* moderate or severe renal impairment: serum creatinine > 1.5 x upper limit of normal (ULN);
* hypersensitivity to any drug of the study regimen;
* unwilling or unable to comply with the protocol for the duration of the study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
2-year survival rate | up to 4 years

SECONDARY OUTCOMES:
Overall response rate | up to 2 years
R0 resection rate | up to 2 years
Operative mortality rate | up to 2 years
in-hospital mortality rate | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guoli Li, M.D., Study Chair — Jinlin Hospital
Locations (1):
- Research institue of general surgery, Jinling hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Xiang XS, Su Y, Li GL, Ma L, Zhou CS, Ma RF. Phase II Study of Preoperative Intra-Arterial Epirubicin, Etoposide, and Oxaliplatin Combined with Oral S-1 Chemotherapy for the Treatment of Borrmann Type 4 Gastric Cancer. J Gastric Cancer. 2020 Dec;20(4):395-407. doi: 10.5230/jgc.2020.20.e40. Epub 2020 Dec 29. PMID 33425441